CLINICAL TRIAL: NCT04036591
Title: Use Of The "Acute Bronchiolitis Severity Scale" In Infants With Acute Respiratory Infection Susceptible To Outpatient Respiratory PhysiotherapyTreatment
Brief Title: Use Of The ABSS In Infants With ARIS Treated With Outpatient Respiratory Physiotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FisioRespiración (Other)
Collaborators: Neumomadrid (Unknown); Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Beatriz Simón Rodríguez, FisioRespiración CEO and physiotherapist, FisioRespiración
Other Study IDs: 19/058-E_TFM
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Acute Disease Respiratory
Keywords: Clinical scale; infant; respiratory therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children under 24 months with ARIS
  Interventions: Diagnostic Test: Acute Bronchiolitis Severity Scale (ABSS)

INTERVENTIONS:
Diagnostic Test: Acute Bronchiolitis Severity Scale (ABSS) — All infants will be assessed using the Acute Bronchiolitis Severity Scale (ABSS) before and after being treated by experienced physiotherapists using the prolonged slow expiration technique and provoqued cough. Before the application of these techniques a retrograde rhinopharyngeal unclogging will be performed in order to clean the nasopharynx.
  Other Names: Chest Physiotherapy

SUMMARY:
Background. Acute respiratory infections in childhood have high incidence and morbimortality rates, generating significant sanitary and social costs. Due to its diversity of manifestations and clinical forms, the degree of severity varies widely.

Published acute respiratory infections assessment severity scales are mainly focused on acute bronchiolitis, but there is no validated scale to evaluate the effects of respiratory physiotherapy in acute respiratory infections in children.

Objective. To study the usefulness of the Acute Bronchiolitis Severity Scale to assess children under 24 months suffering from acute respiratory infections susceptible to receive outpatient respiratory physiotherapy treatment.

Methods. Pre-post assessment descriptive study using the Acute Bronchiolitis Severity Scale. Children under 24 months suffering from acute respiratory infection will be evaluated during the first outpatient respiratory physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Under 24 months
* ARIS diagnosed
* Medical indication of respiratory physiotherapy
* Evaluated during the first outpatient respiratory physiotherapy treatment

Exclusion Criteria:

* Chronic desease
* ABSS ≥ 7
* Temperature≥ 38ºC
* Stridor
* Expiratory groan
* Sternal sinking
* Any sign or symptom indicative of need for urgent medical evaluation

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children who attend to FisioRespiración (Private respiratory physiotherapy unit in Madrid) to receive outpatient respiratory physiotherapy treatment and meet the inclusion/exclusion criteria will be selected until reaching the sample.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Usefulness of Acute Bronchiolitis Severity Score (ABSS) to asses children under 24 months suffering from acute respiratory infection susceptible to receive outpatient respiratory physiotherapy treatment. | Through study completion, an average of 2 years.
  Physiotherapists will use the Acute Bronchiolitis Severity Score (ABSS) to assess severity of infection pre and post treatment. After several assessments each one of them will inform about the usefulness and aplicability of the scale in outpatient respiratory physiotherapy treatment by filling in a likert scale (usefulness, aplicability, simplicity, time required...)
Immediate effectiveness of outpatient respiratory physiotherapy treatment. | Measurements will be taken during the outpatient respiratory physiotherapy treatment, 1 hour approximately. Pre treatment data will be collected before starting the treatment and post data 5 minutes after finishing the last manouver.
  Change from baseline in the Acute Bronchiolitis Severity Score (ABSS) punctuation at the end of outpatient respiratory physiotherapy treatment (pre-post treatment measurement of the scale).
  The ABSS is a validated scale in a Spanish population that combines the evaluation of heart and respiratory rate, wheezings, crackles, respiratory effort and inspiration/exhalation ratio. It has three levels of severity: mild (0 to 4 points), moderate (5 to 9) and severe (10 to 13).

CONTACTS AND LOCATIONS:
Locations (1):
- FisioRespiración, Madrid, Spain